CLINICAL TRIAL: NCT01001702
Title: An Open- Label Rollover Study for Subjects With Schizophrenia Completing ABILIFY® (Aripiprazole) Clinical Study 31-03-241
Brief Title: Oral Aripiprazole Open-Label Rollover Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31-05-243
Record Dates: First submitted 2009-10-22; First posted 2009-10-27 (Estimated); Results first posted 2013-09-27 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-07

CONDITIONS: Schizophrenia
Keywords: Open Label; Aripiprazole
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

ARMS (1):
- Oral Aripiprazole (Experimental): Flexible dose of oral aripiprazole between 5 mg and 30 mg once daily for 72 months.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Flexible dose between 5 mg and 30 mg Aripiprazole tablets.
  Other Names: ABILIFY®

SUMMARY:
The purpose of this study is to test the long-term safety and tolerability of oral aripiprazole in adolescent patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a confirmed Axis I Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnosis of schizophrenia who must have completed Otsuka study 31-03-241 (NCT00102518) treatment of adolescent subjects with schizophrenia

Exclusion Criteria:

* Patients with a co-morbid serious, uncontrolled systemic illness
* Patients with a significant risk of committing suicide

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2006-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- Argentina (2):
  - Study site, Buenos Aires
  - Study site, Mendoza
- Study site, Split, Croatia
- India (4):
  - Study site, Hyderabad
  - Study site, Ludhiana
  - Study site, Mumbai
  - Study site, Tamilnadu
- Russia (4):
  - Study site, Moscow
  - Study site, Rostov-on-Don
  - Study site, Saint Petersburg
  - Study site, Yaroslavl
- Serbia (2):
  - Study site, Belgrade
  - Study site, Novi Sad
- Ukraine (2):
  - Study site, Kharkiv
  - Study site, Kiev

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An open-label rollover study for participants who completed study 31-03-241 (NCT00102518). The withdrawal criteria for this open label rollover study was completion by 31 December 2012 (or if Month 72 occurred within 6 months of this date) or if there was commercial availability.
Period: Overall Study
Arm/Group | Oral Aripiprazole
Started | 85
Completed | 13
Not Completed | 72
Not completed — Lost to Follow-up | 7
Not completed — Adverse Event | 7
Not completed — Sponsor Discontinued Study | 4
Not completed — Subject met Withdrawal Criteria | 22
Not completed — Investigator withdrew Subject | 10
Not completed — Withdrawal by Subject | 19
Not completed — Lack of Efficacy per Investigator | 3

BASELINE CHARACTERISTICS:
Arm/Group | Oral Aripiprazole
Number analyzed (Participants) | 85
Age Continuous [Mean (Standard Deviation); unit: years] | 16.29 (1.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Discontinuation Due to AEs and Deaths
Description: An AE was defined as any new medical problem, or exacerbation of an existing problem, experienced by a subject. Change in clinical relevance (severity increased) was entered as a new AE in the current trial. Abnormal laboratory test findings were considered AEs if, in the opinion of the investigator, they represented an abnormal (clinically significant) change from baseline for that individual subject.
  An AE was considered serious if it was fatal; life-threatening; persistently or significantly disabling or incapacitating; required in-patient hospitalization or prolonged hospitalization; a congenital anomaly/birth defect; or other medically significant event that, based upon appropriate medical judgment, may have jeopardized the subject and may have required medical or surgical intervention.
  Additional information about Adverse Events can be found in the Adverse Event section.
Time Frame: Up to 72 months
Population: Safety population included all participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Oral Aripiprazole
Number analyzed (Participants) | 85
Participants
  AEs | 61
  SAEs | 11
  Discontinuation due to AEs | 7
  Death | 1

2. Secondary Outcome: Change From Baseline in Clinical Global Impression Severity of Illness (CGI-S) Score
Description: The rater or investigator answered the following question:
  "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" Response choices included: 0=not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients. A negative change from Baseline indicated improvement
Time Frame: Baseline, Last Visit (Up to 72 Months)
Population: Participants with baseline assessment and at least one post-baseline measurement for analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Aripiprazole
Number analyzed (Participants) | 84
Score on a scale | -0.26 (1.07)

3. Secondary Outcome: Number of Participants With Clinical Significant Laboratory Tests
Description: Blood was collected for Fasting clinical laboratory tests (serum chemistry and hematology) at Baseline, Months 12, 24, 36, 48, 60, and 72 and were analyzed at a central laboratory.
  Clinically significant values are defined as the following:
  Bilirubin, total ≥ 2.0 mg/dL. Creatine phosphokinase > 500 U/L for participants 13-17 years or 3 times the upper limit of normal for participants ≥ 18 years [Reference Range (0 to 190 IU/L (females) and 0 to 235 IU/L (males)].
  Eosinophils ≥ 10 %. Hematocrit < 30 % for participants 13-17 years old or ≥ 18 year old participants female ≤ 32 % and a 3 point decrease from baseline or male ≤ 37 % and a 3 point decrease from baseline.
  Hemoglobin female ≤ 9.5 g/dL or male ≤ 11.5 g/dL. Prolactin > 1 times the upper limit of normal [Reference range: 2 to 18 ng/mL (males) and 3 to 30 ng/mL (females)].
Time Frame: Baseline, Up to 72 Months
Population: Participants with at least one post-baseline numeric result for the given laboratory test are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Oral Aripiprazole
Number analyzed (Participants) | 79
Participants
  Bilirubin, total (mg/dL) | 7
  Creatine phosphokinase (CPK), total (IU/L) | 6
  Eosinophils (%) | 5
  Hematocrit (%) | 5
  Hemoglobin (g/dL) | 3
  Prolactin (ng/mL) | 3

4. Secondary Outcome: Number of Participants With Clinically Significant Heart Rate
Description: Heart rate was measured at Baseline and at each visit supine (lying on the back) and standing. A heart rate increase is an increase of ≥ 15 beats per minute (bpm) compared to Baseline. A heart rate decrease is a decrease of ≥ 15 bpm compared to Baseline.
Time Frame: Baseline, Up to 72 months
Population: Participants with baseline assessment and at least one post-baseline numeric result for the given parameter.
Measure: Number; unit: Participants
Arm/Group | Oral Aripiprazole
Number analyzed (Participants) | 84
Participants
  Supine Heart Rate Increase | 0
  Supine Heart Rate Decrease | 0
  Standing Heart Rate Increase | 1
  Standing Heart Rate Decrease | 0

5. Secondary Outcome: Number of Participants With Clinically Significant Blood Pressure
Description: Systolic and Diastolic blood pressure was measured at Baseline and at all visits supine (lying on the back) and standing.
  Systolic increase was an increase of ≥ 20 mm Hg compared to Baseline and systolic decrease was a decrease of ≥ 20 mm Hg compared to Baseline.
  A diastolic increase was an increase of ≥ 15 mm Hg compared to Baseline and a diastolic decrease was a decrease of ≥ 15 mm Hg compared to Baseline.
Time Frame: Baseline, Up to 72 months
Population: Participants with baseline assessment and at least one post-baseline numeric result for the given parameter.
Measure: Number; unit: Participants
Arm/Group | Oral Aripiprazole
Number analyzed (Participants) | 84
Participants
  Supine Systolic Blood Pressure Increase | 4
  Supine Systolic Blood Pressure Decrease | 3
  Standing Systolic Blood Pressure Increase | 5
  Standing Systolic Blood Pressure Decrease | 2
  Supine Diastolic Blood Pressure Increase | 5
  Supine Diastolic Blood Pressure Decrease | 0
  Standing Diastolic Blood Pressure Increase | 5
  Standing Diastolic Blood Pressure Decrease | 0

6. Secondary Outcome: Number of Participants With Clinically Abnormal Changes in Electrocardiograms (ECGs) Evaluations
Description: A 12-lead ECG was recorded at Baseline, Months 6, 12, 24, 36, 48, 60 and 72. Three readings taken 5 minutes were read by a central ECG reading service and averaged.
  Clinically significant ECGs were defined as:
  Sinus Bradycardia: ≤ 50 beats per minute (bpm), decrease of ≥ 15 bpm from Baseline.
  Supraventricular premature beat: ≥ 2 per 10 seconds, increase from Baseline. Ventricular premature beat: ≥ 1 per 10 seconds, increase from Baseline. Right bundle branch block: present. Other intraventricular block: QRS ≥ 0.10 seconds for age 13-17 years or QRS ≥ 0.11 seconds for age ≥ 18 years, an increase of ≥ 0.02 seconds from Baseline.
  Symmetrical T-wave inversion: present. QTcB (QT interval corrected Bazett's formula), QTcF (QT interval corrected Fridericia's formula), QTcN (QT corrected FDA Neuropharmacology Division formula), QTcE (QT corrected fractional exponent correction method: ≥ 420 msec for age 13-17 years or ≥ 450 msec for age ≥ 18 years, ≥ 10 % increase from Baseline.
Time Frame: Baseline, Up to 72 months
Population: Participants with at least one post-baseline numeric result for the given parameter.
Measure: Number; unit: Participants
Arm/Group | Oral Aripiprazole
Number analyzed (Participants) | 82
Participants
  Sinus bradycardia | 7
  Supraventricular premature beat | 6
  Ventricular premature beat | 1
  Right bundle branch block | 1
  Other intraventricular block | 5
  Symmetrical T-wave inversion | 1
  QTcB | 9
  QTcF | 4
  QTcN | 6
  QTcE | 5

7. Secondary Outcome: Number of Participants Showing Significant Weight Gain or Loss
Description: Weight was measured at Baseline, Months 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, and 72. A clinically significant weight gain was defined as a ≥ 7 % increase from Baseline. A clinically significant Weight loss was defined as a ≥ 7% decrease from Baseline.
Time Frame: Baseline, Up to 72 months
Population: Participants with baseline assessment and at least one post-baseline numeric result for the given parameter.
Measure: Number; unit: Participants
Arm/Group | Oral Aripiprazole
Number analyzed (Participants) | 82
Participants
  Weight Gain | 37
  Weight Loss | 4

8. Secondary Outcome: Number of Participants Experiencing Suicidal Ideation or Suicidal Behavior Based on Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS consisted of a baseline evaluation (completed at the first scheduled visit upon approval of protocol Amendment 3) that assessed the lifetime experience of the participant with suicide events and suicidal ideation and a post-baseline evaluation at each visit that focused on suicidality since the last trial visit. Some questions are yes/no and some are on a scale of 1 (low severity) to 5 (high severity). The number of participants experiencing suicidal ideation or suicidal behavior is reported.
Time Frame: Baseline, Up to 72 months
Population: All participants with available assessment.
Measure: Number; unit: Participants
Arm/Group | Oral Aripiprazole
Number analyzed (Participants) | 14
Participants | 0

ADVERSE EVENTS:
Arm/Group | Oral Aripiprazole
Serious Adverse Events (participants affected / at risk) | 11/85
Other Adverse Events (participants affected / at risk) | 45/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Aripiprazole (N=85)
Pneumonia bacterial (Infections and infestations) | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1
Psychomotor hyperactivity (Nervous system disorders) | 1
Aggression (Psychiatric disorders) | 1
Impulsive behaviour (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 2
Suicide attempt (Psychiatric disorders) | 3
Social stay hospitalisation (Social circumstances) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Aripiprazole (N=85)
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 7
Pain (General disorders) | 7
Influenza (Infections and infestations) | 9
Nasopharyngitis (Infections and infestations) | 6
Weight increased (Investigations) | 9
Decreased appetite (Metabolism and nutrition disorders) | 5
Headache (Nervous system disorders) | 13
Somnolence (Nervous system disorders) | 5
Anxiety (Psychiatric disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Pyrexia (General disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No